CLINICAL TRIAL: NCT05156801
Title: Efficacy of the ArchSinus, NasoPore and the Propel Stent in Preventing Post-Surgical Middle Turbinate Lateralization and Improving the Symptomatic Outcomes; Randomized, Blinded, Comparative Study
Brief Title: Efficacy of ArchSinus, NasoPore & Propel to Prevent Post-Surgical MT Lateralization and Improve Symptomatic Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: STS Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 461008P
Record Dates: First submitted 2021-11-29; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Intervention Model Description: 50 chronic rhinosinusitis patients, that met the inclusion criteria will undergo randomization into ArchSinus / Propel or ArchSinus / NasoPore implantation group. Comparative treatment sides will be randomly assigned; 13 subjects will be assigned to ArchSinus (right)/ Propel (left); 12 subjects will be assigned to ArchSinus (left)/ Propel (right); 12 subjects will be assigned to ArchSinus (right)/ NasoPore (left); 13 subjects will be assigned to ArchSinus (left)/ NasoPore (right) groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Primary objective will be analyzed using nasal video endoscopy and a CT scan, by an external experts in a blinded fashion. Secondary objective will be analyzed using side-specific SNOT-22 questioner, subjects will be blinded to the treatment type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ArchSinus stent (Experimental): Post-FESS implantation of the study device (ArchSinus) into ethmoid sinus cavity
  Interventions: Device: ArchSinus stent
- Propel stent (Active Comparator): Post-FESS implantation of the comparator device (Propel) into ethmoid sinus cavity.
  Interventions: Device: ArchSinus stent
- NasoPore packing (Active Comparator): Post-FESS implantation of the comparator device (NasoPore) into ethmoid sinus cavity.
  Interventions: Device: ArchSinus stent

INTERVENTIONS:
Device: ArchSinus stent — Post FESS unilateral placement of the ArchSinus stent into the randomized ethmoid sinus cavity.
  Other Names: Composite Removable Sinus Stent System

SUMMARY:
This is a multi-center, randomized, single-blinded comparative 3-arm clinical study. This clinical study is designed to compare the efficacy of the ArchSinus stent to the Propel stent (Intersect ENT), and to NasoPore (Stryker) in preventing post-FESS middle turbinate lateralization 3 weeks, 6 weeks, 3 months and 12 months post FESS.

DETAILED DESCRIPTION:
50 chronic rhinosinusitis patients, that met the inclusion criteria will undergo bilateral FESS and subsequent bilateral placement of the ArchSinus into the randomized ethmoid sinus cavity and NasoPore / Propel into the other ethmoid sinus cavity. Comparative treatment sides will be randomly assigned; 50 sinuses treated with ArchSinus stent, 25 sinus treated with Propel stent, 25 sinuses treated with Nasopore. Standard Propel implant and 4cm whole NasoPore will be used.

ArchSinus stent will be removed 2 weeks (13-15 days) post FESS. Propel will be removed as necessary 2 weeks (13-15 days) post FESS. NasoPore arm will be debrided as necessary 2 weeks (13-15 days) post-FESS. Prior to removal / debridement procedures, the patients will be blindfolded, to keep them blinded for the treatment type on each side of their nose.

All patients will be followed up at 2, 6 and 12 weeks and 12 months post FESS and examined endoscopically. The endoscopic videos will be analyzed by independent pannel of 3 ENT surgeons, blinded to the treatment type, to assess middle turbinate lateralization on a 4-point scale.

CT scan will be performed pre-FESS and 12 weeks after the operation, to assess middle turbinate lateralization, as demonstrated by percent change in middle meatus (MM) area pre-FESS and 12 weeks after the surgery. Inflammatory mucosal thickening will be quantified using the Zinreich staging system. CT scans will be analyzed blindly by Medical Metrics Inc.

Symptomatic improvement will be analyzed weekly within 3 months follow up, using Side-specific Nasal SNOT-22 questioner.

Patient symptomatic relief during the implantation time will be analyzed 2 weeks post FESS, with Side-specific Nasal SNOT-22 questioner.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis defined as symptomatic inflammation of the sinuses of at least 12 consecutive weeks duration despite medical management
* CT scan examination with a minimum Zinreich score of 5 prior to study entry
* Less than 2-point Zinreich score difference between two sides
* Primary FESS including bilateral total ethmoidectomy; symmetrical uncinate process reduction

Exclusion Criteria:

* Inferior turbinectomy, reduction or outfracture
* Polyp grade ˃ 4 bilaterally on Lildholdt's scale (1-3)
* Concha bullosa
* Severe nasal septal deviation at the level of OMC
* Sinonasal tumors
* FESS including asymmetrical resection of the middle turbinate
* Known allergy to nickel
* Known polyurethane induced dermatitis
* Oral steroid-dependent condition
* Momometasone furoate intolerance
* Known hypersensitivity to lactide, glycolide or caprolactone copolymers.
* Glaucoma or cataract
* History of immune deficiency
* Cystic fibrosis
* Pregnant or lactating female
* Acute sinus inflammation
* Coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Middle turbinate lateralization 12 week post FESS (based CT scan) | 12 weeks post FESS
  The primary objective is to compare the efficacy of the ArchSinus to Propel stent (Intersect ENT), to prevent post-FESS middle turbinate lateralization, 12 weeks post-FESS, based on CT scan.

SECONDARY OUTCOMES:
Middle turbinate lateralization 12 week post FESS (based video endoscopy) | 12 weeks post FESS
  The secondary objective (1) is to compare the efficacy of the ArchSinus to the Propel stent (Intersect ENT), ), to prevent post-FESS middle turbinate lateralization, 12 weeks post-FESS, based on video endoscopy on a 4-point scale.
Symptomatic outcomes within the 3-month post-FESS | 12 weeks post FESS
  The secondary objective (2) is to compare the efficacy of the ArchSinus to the Propel stent (Intersect ENT) in improving the symptomatic outcomes based on side-specific SNOT-22 questioner, within the 3-month follow-up.

OTHER OUTCOMES:
Re-stenosis rate 6 weeks post FESS (based video endoscopy) | 6 weeks post FESS
  (1) Compare re-stenosis rate in ArchSinus / Propel / NasoPore implanted sinuses assessed on a 1 to 4 scale based on nasal endoscopy at week 6
symptomatic relief 2 weeks post FESS | 2 weeks post FESS
  Compare symptomatic relief in ArchSinus / Propel / NasoPore implanted sinuses, based side - specific Nasal SNOT-22 score 2 weeks post-FESS.
Removal time | 2 weeks post FESS
  Compare ArchSinus and Propel removal time
Inflammatory mucosal thickening | 12 weeks post FESS
  Compare % change of inflammatory mucosal thickening 12 weeks post FESS in ArchSinus / Propel / NasoPore implanted sinuses
Re-stenosis rate 12 months post FESS | 12 months post FESS
  Compare re-stenosis rate in ArchSinus / Propel / NasoPore implanted sinuses assessed on a 1 to 4 scale based on nasal endoscopy 12 months post FESS.